CLINICAL TRIAL: NCT03292614
Title: Measurement of Refraction Following Cataract Surgery With Implantation of MICS Intraocular Lens LS313 MF30, Oculentis Berlin
Brief Title: Measurement of Refractive SE Following Implantation of LS313 MF30 IOL
Status: Completed | Type: Observational
Sponsor: Dietrich-Bonhoeffer-Klinikum (Industry)
Responsible Party: Sponsor
Other Study IDs: STI 02/17
Record Dates: First submitted 2017-09-21; First posted 2017-09-25 (Actual); Results first posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-08

CONDITIONS: Refractive Errors
Keywords: Multifocal Intraocular Lens; Postoperative Measurements of refraction
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multifocal intraocular lens implantation: Patients who have undergone a cataract surgery with implantation of a multifocal intraocular lens LS313 MF30, Oculentis Berlin, will be invited for Measurements of the postoperative refraction
  Interventions: Diagnostic Test: Measurements of the postoperative refraction

INTERVENTIONS:
Diagnostic Test: Measurements of the postoperative refraction — The Measurements of the postoperative refraction will be performed with the following devices:
  Autorefractor Keratometers:
  Mod. ARK-760A (NIDEK CO,LTD, Gamagõri, Japan /OCULUS, Wetzlar, Germany), Mod. ARK-560A (NIDEK CO,LTD, Gamagõri, Japan /OCULUS, Wetzlar, Germany) KR-1W (TOPCON, Willich, Germany) KR-800s (TOPCON, Willich, Germany)
  Manual Refractometer:
  Eye refractometer PR 60 or PR 50 (Rodenstock, Munich),
  Test device:
  iTrace (TraceyTechnologies, Houston, Texas, USA),
  Phoropter (Block-Optic, Model 11625B) Determination of subjective refraction for distance and near (reading distance)

SUMMARY:
This Study determines the most precise method for measuring post-operative refraction following implantation of the asymmetric multifocal LS-313 MF30 comparing the results of Refraction of the different Autorefractor Keratometers with the subjective measurements for distance and near.

DETAILED DESCRIPTION:
This is a post market study without invasive interventions. The patients have been treated with cataract surgery and MIOL Implantation at least 3 months ago. They will be invited for only one follow up visit to measure the postoperative refraction with different Autorefractor-Keratometers, a Manual Refractometer, the test device "iTrace" and with determination of the subjective refraction for distance and near with the appropriate corrections at the Department of Ophthalmology in Neubrandenburg, Germany.

ELIGIBILITY:
Inclusion Criteria:

Patients after cataract surgery with implantation of the MICS-IOL LS-313 MF30 postoperative clear cornea willing to participate in the study

Exclusion Criteria:

significant corneal opacities, history of keratoplasty, Anterior capsule phimosis, posterior capsular opacification if patients refuse Nd:YAG laser treatment of the secondary cataract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: up to 100 eyes
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Hoeh, MD, FEBO, Principal Investigator — Department of Ophthalmology, Neubrandenburg, Germany; Vitaliy Klishko, Study Chair — Department of Ophthalmology, Neubrandenburg, Germany
Locations (1):
- Dietrich-Bonhoeffer-Klinikum, Neubrandenburg, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in ophthalmological journals (Individual participant date will not be provided).

REFERENCES:
- [Background] Kretz FT, Linz K, Mueller M, Gerl M, Koss MJ, Gerl RH, Auffarth GU. [Refraction after Implantation of Multifocal and Presbyopia-Correcting Intraocular Lenses]. Klin Monbl Augenheilkd. 2015 Aug;232(8):953-6. doi: 10.1055/s-0035-1545832. Epub 2015 Apr 30. German. PMID 25927177
- [Background] Munoz G, Albarran-Diego C, Sakla HF. Validity of autorefraction after cataract surgery with multifocal ReZoom intraocular lens implantation. J Cataract Refract Surg. 2007 Sep;33(9):1573-8. doi: 10.1016/j.jcrs.2007.05.024. PMID 17720072
- [Background] Bissen-Miyajima H, Minami K, Yoshino M, Nishimura M, Oki S. Autorefraction after implantation of diffractive multifocal intraocular lenses. J Cataract Refract Surg. 2010 Apr;36(4):553-6. doi: 10.1016/j.jcrs.2009.10.047. PMID 20362844
- [Background] van der Linden JW, Vrijman V, Al-Saady R, van der Meulen IJ, Mourits MP, Lapid-Gortzak R. Autorefraction versus subjective refraction in a radially asymmetric multifocal intraocular lens. Acta Ophthalmol. 2014 Dec;92(8):764-8. doi: 10.1111/aos.12410. Epub 2014 Apr 27. PMID 24767468
- [Background] Munoz G, Albarran-Diego C, Sakla HF. Autorefraction after multifocal IOLs. Ophthalmology. 2007 Nov;114(11):2100. doi: 10.1016/j.ophtha.2007.05.049. No abstract available. PMID 17980752

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Multifocal Intraocular Lens Implantation
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Multifocal Intraocular Lens Implantation
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.84 (8.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 25

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of the Most Precise Method for Measuring Post-operative Refraction Following Implantation of the Asymmetric Multifocal LS-313 MF30
Description: After the implantation of the LS 313 MF30 (a refractive, asymmetrical, multifocal intraocular lens), the most reliable refraction method so far has been the subjective determination of far and near refraction.
  A faster and widespread method is the measurement with auto-refractometers (KR-1W (TOPCON), KR-800s (TOPCON), ARK-560 (NIDEK), ARK-760A (NIDEK)) or manual refractometers (PR60/50 (Rodenstock)).
  KR-1W, KR-800s, ARK-560A, ARK-760A only allow a central measurement without separate measurement of the two optical zones.
  The manual refractometer PR60/50 (Rodenstock) is able to separately measure the different focal points of the multifocal lens using a light cone with 3 mm diameter.
  The test device iTrace (TraceyTechnologies): is also able to separately measure the different focal points of the multifocal lens, but uses a light cone with a diameter of about 1 mm.
  The results of all refractometers are compared with the subjective refraction.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: diopter
Arm/Group | Multifocal Intraocular Lens Implantation
Number analyzed (Participants) | 25
diopter
  subjective Refraction | 0.36 (0.65)
  iTrace | 0.27 (0.64)
  KR-W1 | -0.81 (0.59)
  KR-800s | -0.78 (0.73)
  ARK-760A | -0.73 (0.59)
  ARK-560A | -0.76 (0.63)
  PR60/50 | -0.18 (0.43)

ADVERSE EVENTS:
Time Frame: 1 month
Description: Adverse events that may occur in the course of this study are glare sensitivity, allergic reaction, continuous dilation over 2 to 3 days (in Mydriasis) or accident on the way to the investigations.
Arm/Group | Multifocal Intraocular Lens Implantation
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/14/NCT03292614/Prot_000.pdf